CLINICAL TRIAL: NCT06396325
Title: A Registry-Based Parallel Group Randomized-Controlled Trial of an Upper Limb Exergaming Intervention for Children and Adolescents With Spinal Muscular Atrophy, With an Optional Open-Label Extension
Brief Title: A Registry Based Randomized-Controlled Trial of an Upper Limb Exergaming Intervention for Children and Adolescents With Spinal Muscular Atrophy
Acronym: INFORM SMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maryam Oskoui, MD, MSc, FRCPC, FAAN (Other)
Responsible Party: Sponsor-Investigator, Maryam Oskoui, MD, MSc, FRCPC, FAAN, Full Professor, Department of Pediatrics and Neurology & Neurosurgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-37-2022-7289
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; rehabilitation; Exergaming; Pediatrics; Randomized-controlled trial
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exergaming Intervention for 8 Weeks (Experimental): Extension Phase: Participants randomized ot the intervention arm will play Tales from the Magic Keep at home for the 8 week open-label extension phase
  Interventions: Other: Tales from the Magic Keep™
- Usual Care for 8 weeks. (Active Comparator): Extension Phase: Participants randomized to waitlist usual care will play Tales from the Magic Keep at home for the 8 week open-label extension phase
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Tales from the Magic Keep™ — Exergame targeting upper limb and trunk movement designed for use on the Microsoft Azure Kinect Dose: At least 3 times a week for 20 minutes over 8 weeks (8 hours total) Continue with regularly accessed physical activities and rehabilitation services
  Arms: Exergaming Intervention for 8 Weeks
Other: Usual Care — Continue with regularly accessed physical activities and rehabilitation services
  Arms: Usual Care for 8 weeks.

SUMMARY:
This is a multisite randomized controlled registry-based trial to evaluate the efficacy of an 8-week home-based exergaming intervention as compared to usual care on occupational satisfaction of children and youth (8-18 years old age) with spinal muscular atrophy (SMA).

DETAILED DESCRIPTION:
This multisite randomized controlled registry-based trial will evaluate the efficacy of a home-based exergaming intervention, as compared to usual care, on occupational satisfaction of children and youth (aged 8-18 years old) with SMA. Participants in the intervention arm will play the exergame, Tales from the Magic Keep™ on the Azure Kinect platform, 3 times per week, for at least 20 minutes, over 8 weeks (total 8 hours), and continue to access their regular physical activities and rehabilitation services. Those in the usual care arm will continue to access their regular physical activities and rehabilitation services. Occupational satisfaction will be assessed using the Canadian Occupational Performance Measure (COPM) at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed genetic diagnosis of 5q SMA
* Age at screening: Aged 8-18 years old
* Participant is able to stay seated independently without support for at least 10 seconds
* Participants has a score of at least 2 points in entry item A of the RULM (i.e., "Can raise 1 or 2 hands to the mouth but cannot raise a 200 g weight in it to the mouth")
* Treated with disease-modifying therapy
* Signed ICF

Exclusion Criteria:

* Inability to comply with study procedures according to the site investigator, prior to randomization
* Severe scoliosis or contractures that would interfere with gameplay or with successful completion of functional assessments, as confirmed by the clinical evaluator
* Planned orthopedic surgery 6 months prior to or throughout intervention and follow-up period (16 weeks post randomization)
* Inability to read in English or French

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with occupational performance | Baseline to 16 weeks
  Canadian Occupational Performance Measure (COPM) Satisfaction

SECONDARY OUTCOMES:
Self-reported fatigue | Baseline to 16 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS-SF)
Independence performing activities of daily living | Baseline to 16 weeks
  SMA Independence Scale (SMAIS)
Upper limb motor activity | Baseline to 16 weeks
  Median and 99th percentile of upper limb rotational effort and vertical wrist acceleration derived from data captured by the Syde wearable device

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Oskoui, Principal Investigator — McGill University; Danielle Levac, Principal Investigator — Université de Montréal
Locations (5):
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Services, Halifax, Nova Scotia
  - Hospital for SickKids, Toronto, Ontario
  - Centre de readaptation Marie-Enfant, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No